CLINICAL TRIAL: NCT00215137
Title: Pilot Study to Evaluate Escitalopram in Obsessive-compulsive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00013150; 5731-04-4R0 (Other: Duke legacy protocol number)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Results first posted 2013-10-29 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2013-08

CONDITIONS: OCD
Keywords: OCD; SSRI; escitalopram; relapse
MeSH Terms: conditions — Recurrence | interventions — Escitalopram; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Open Label Escitalopram 10-20 mg/daily (Experimental): Fourteen patients who met criteria for the study were enrolled in the open-label phase. Thirteen of these patients completed the open-label phase, while one patient was terminated early due to side effects.
  Interventions: Drug: escitalopram
- Randomizationn Placebo 10-20 mg daily (Placebo Comparator): Of the thirteen patients who completed the open label part of the trial, twelve demonstrated at least minimal improvement (CGI-I < 3) and agreed to continue with the randomized, double-blind phase. These patients were randomized to escitalopram (n=5) or placebo (n=7).
  Interventions: Drug: Placebo ( sugar pill)
- Randomization Escitalopram 10-20 mg/daily (Active Comparator): Of the thirteen patients who completed the open label part of the trial, twelve demonstrated at least minimal improvement (CGI-I < 3) and agreed to continue with the randomized, double-blind phase. These patients were randomized to escitalopram (n=5) or placebo (n=7).
  Interventions: Drug: escitalopram

INTERVENTIONS:
Drug: escitalopram — Open label Treatment: Escitalopram 10 mg/day for 1 week and then 20 mg /day for 7 weeks. Double Blind Treatment: Escitalopram 20 mg/day.
  Other Names: Lexapro
  Arms: Open Label Escitalopram 10-20 mg/daily; Randomization Escitalopram 10-20 mg/daily
Drug: Placebo ( sugar pill) — Placebo Comparator in double.blind phase.
  Other Names: Placebo
  Arms: Randomizationn Placebo 10-20 mg daily

SUMMARY:
This study will determine the safety and effectiveness of escitalopram (Lexapro)in treating obsessive-compulsive disorder (OCD) symptoms.

DETAILED DESCRIPTION:
OCD is a chronic and disabling disorder for which Selective Serotonin Reuptake Inhibitor(SSRI) drugs can be effective. The purpose of this study is to evaluate the effects of an SSRI, escitalopram, in OCD patients.

This study will last 16 weeks and will comprise 2 phases. Phase 1 is an open label in which all participants will receive daily escitalopram for 8 weeks. Those who have responded to treatment at the end of the 8 weeks will be randomly assigned to either continue or discontinue their treatment for an additional 8 weeks. Those who do not respond to treatment at the end of Phase 1 will discontinue the study and be offered three free visits with a study clinician or referred elsewhere for treatment, based on the their preference. Study visits are made at baseline, and at Weeks 1, 2, 4, and 8 in Phase 1 and Weeks 12 and 16 in Phase 2.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of OCD
* A minimum score of 16 on the Yale Brown Obsessive-Compulsive Scale (YBOCS) at both the screening and baseline visits

Exclusion Criteria:

* Lifetime history of psychosis or cognitive dysfunction due to a general medical condition or substance use
* A primary diagnosis of another Axis I psychiatric disorder
* Alcohol or other substance abuse or dependence within the last 6 months
* Unstable medical condition
* Clinically significant laboratory abnormality
* Failure of a previous 10-week trial of citalopram of at least 40 mg/day or escitalopram 20 mg/day
* Active suicidality
* History of violent behavior in the past year or current risk of serious violence
* A history of sensitivity to citalopram or escitalopram
* Use of other investigational drugs within 30 days of baseline or other psychotropic drugs or herbs within 14 days of baseline (28 days for fluoxetine)
* Need for concurrent psychotherapeutic intervention
* Pregnant or lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2004-10; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wei M. Zhang, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Result] C. Joseph Wang, M.D., Ph.D.; Jonathan R. Davidson, M.D.; Kathryn M. Connor, M.D.;Weihui Li1, M.D.,Ph.D. and Wei Zhang, M.D., Ph.D. Unpublished Manuscript

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label Escitalopram: Fourteen patients who met criteria for the study were enrolled in the open-label phase. Thirteen of these patients completed the open-label phase, while one patient was terminated early due to side effects.
- Randomization Placebo; Randomization Escitalopram: Of the thirteen patients who completed the open label part of the trial, twelve demonstrated at least minimal improvement (CGI-I < 3) and agreed to continue with the randomized, double-blind phase. These patients were randomized to escitalopram (n=5) or placebo (n=7).
Period: Open Label Escitalopram
Arm/Group | Open Label Escitalopram | Randomization Placebo | Randomization Escitalopram
Started | 14 | 0 | 0
Completed | 13 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Period: Randomization Period
Arm/Group | Open Label Escitalopram | Randomization Placebo | Randomization Escitalopram
Started | 0 | 7 | 5
Completed | 0 | 5 | 5
Not Completed | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Only the open label treatment phase is being reported per reviewer's instructions. The other arms are for the second phase of the study.
Arm/Group | Open Label Escitalopram
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.14 (13.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Yale Brown Obsessive Compulsive Scale
Description: The Yale Brown Obsessive Compulsive Scale (YBOCS) is a clinician administered measure of the severity of obsessive compulsive disorder(OCD). Higher scores indicate a greater severity of OCD symptoms. The score can range from a minimum of zero to a maximum of forty.
Time Frame: Open Label Phase Baseline,Randomization Phase Baseline or Beginning
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Open Label Escitalopram: Fourteen patients who met criteria for the study were enrolled in the open-label phase. Thirteen of these patients completed the open-label phase, while one patient was terminated early due to side effects.Data presented is based on an intent to treat (ITT), last observation carried forward (LOCF) from post baseline sample.
- Randomization Placebo: Of the thirteen patients who completed the open label part of the trial, twelve demonstrated at least minimal improvement (CGI-I < 3) and agreed to continue with the randomized, double-blind phase. These patients were randomized to escitalopram (n=5) or placebo (n=7).Data presented is based on an intent to treat (ITT), last observation carried forward (LOCF) from post beginning of the study phase sample.
- Randomization Escitalopram: Of the thirteen patients who completed the open label part of the trial, twelve demonstrated at least minimal improvement (CGI-I < 3) and agreed to continue with the randomized, double-blind phase. These patients were randomized to escitalopram (n=5) or placebo (n=7).Data presented is based on an intent to treat (ITT), last observation carried forward (LOCF) from beginning of the study phase sample.
Arm/Group | Open Label Escitalopram | Randomization Placebo | Randomization Escitalopram
Number analyzed (Participants) | 14 | 7 | 5
units on a scale
  Beginning of Study Phase | 24.79 (4.48) | 12.71 (6.13) | 16.00 (6.96)
  End of Study Phase | 15.36 (7) | 20.17 (11.57) | 15.8 (7.79)
Statistical Analysis 1: Comparison: Open Label Escitalopram; A Wilcoxon Signed Rank test was performed on the difference between the open label endpoint and baseline YBOCS scores; Test type: Superiority or Other; p = 0.0002, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Randomization Placebo vs Randomization Escitalopram; A Wilcoxon Rank Sum Test was performed on the difference in the pre and post randomization YBOCS scores, using grouping to either escitalopram or placebo as a grouping variable; Test type: Superiority or Other; p = .0417, Wilcoxon Rank Sum Test

ADVERSE EVENTS:
Arm/Group | Open Label Escitalopram | Randomization Placebo | Randomization Escitalopram
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 0/14 | 0/7 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No